CLINICAL TRIAL: NCT01209624
Title: Prospective, Observational Study to Investigate the Long-term Effect of Xalatan® on Intraocular Pressure (IOP) and on Maintenance of Visual Field in Patients With Normal Tension Glaucoma (NTG)
Brief Title: Observational Study of the Long-term Effect of Latanoprost in Normal Tension Glaucoma
Acronym: NTG-X-PERT
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6111135; A6111135
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2010-10-26 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2011-06

CONDITIONS: Low Tension Glaucoma
Keywords: prospective; non-interventional; observational; multi-center; long-term
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the long-term efficacy and safety of latanoprost monotherapy in patients with normal tension glaucoma (NTG) using a prospective, observational design. Visits were scheduled at 6-month intervals for 24 months. Intraocular pressure (IOP), optic nerve head findings, visual field status, and adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

patients with normal-tension glaucoma

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma subjects
Sampling Method: Non-Probability Sample
Enrollment: 902 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111135&StudyName=Observational%20Study%20of%20the%20Long-term%20Effect%20of%20Latanoprost%20in%20Normal%20Tension%20Glaucoma%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this prospective non-interventional study, participants did not actively participate in the study but were observed in general clinical practice by office-based ophthalmologists.
Groups:
- Xalatan®: Once daily as 1 drop (topical application) in the evening
Period: Overall Study
Arm/Group | Xalatan®
Started | 902
Per Protocol Population | 469
Completed | 576
Not Completed | 326
Not completed — Death | 2
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 17
Not completed — Lost to Follow-up | 290
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Xalatan®
Number analyzed (Participants) | 902
Age, Customized [Number; unit: participants]
  < 18 years | 5 (13.1)
  18 to 44 years | 68
  45 to 64 years | 281
  >= 65 years | 528
  unspecified | 20
Sex/Gender, Customized [Number; unit: participants]
  Female | 545
  Male | 347
  Unspecified | 10
Raw Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] — Mean IOP value measured by applanation tonometry or noncontact method; valid range: 8-40 millimeters of mercury (mmHg). Only the IOP reading for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  mmHg | 18.14 (3.62)
Horizontal Cup to Disc Ratio [Mean (Standard Deviation); unit: Ratio] — Mean horizontal cup to disc ratio measured by slit lamp examination to assess progression of glaucoma; calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc). Valid range: 0.1-1.0. Only data for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may be represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  Ratio | 0.53 (0.22)
Vertical Cup to Disc Ratio [Mean (Standard Deviation); unit: Ratio] — Mean vertical cup to disc ratio measured by slit lamp examination to assess progression of glaucoma; calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc). Valid range: 0.1-1.0. Only data for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may be represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  Ratio | 0.56 (0.22)
Rim Area [Mean (Standard Deviation); unit: mm^2] — Rim area (millimeter [mm]2) right and left eye assessed by HRT imaging. Valid range: 0.500 to 1.900 mm2. Only the rim area for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may represent more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  mm^2 | 1.26 (0.30)
Rim Volume [Mean (Standard Deviation); unit: mm^3] — Rim volume (mm3) right and left eye assessed by HRT imaging. Valid range: 0.080 to 0.700 mm3. Only the rim volume for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may be represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  mm^3 | 0.30 (0.14)
Cup Shape Measure [Mean (Standard Deviation); unit: Cup shape measure] — Cup shape measure right and left eye assessed by HRT imaging. Valid range: -0.400 to -0.010. Only the cup shape measure for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may be represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  Cup shape measure | -0.12 (0.09)
Retinal Nerve Fiber Layer Thickness [Mean (Standard Deviation); unit: mm] — Mean retinal nerve fiber layer (RNFL) thickness in millimeters (mm) right and left eye assessed by HRT imaging. Valid range: 0.100 to 0.400 mm. Only the RNFL for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may be represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  mm | 0.21 (0.07)
Optic Disc Hemorrhage [Number; unit: Participants] — Presence of optic disc hemorrhages assessed by slip lamp examination. Only data for eye were treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Participants may be represented in more than 1 category. Results based on participants in PP population with a non-missing response at baseline.
  Participants | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Raw Intraocular Pressure (IOP) by Visit
Description: Mean IOP values measured by applanation tonometry or noncontact method; valid range: 8-40 millimeters of mercury (mmHg). Only the IOP reading for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed. Last visit = last post-baseline visit at which participant provides a value of IOP.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: Per protocol (PP) analysis set: all participants in the Full Analysis Set (at least 1 dose of Xalatan® and 1 post-baseline IOP measurement) who were treated for ≥18 months; had at least BL and 1 post-BL non-missing efficacy assessments for IOP at least 18 months apart; without ametropy at BL; and without additional glaucoma medication during study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
mmHg
  Month 6 | -3.20 (3.11)
  Month 12 | -3.12 (3.35)
  Month 18 | -3.22 (3.52)
  Month 24 | -3.43 (3.51)
  Last Visit | -3.34 (3.59)

2. Primary Outcome: Number of Participants With a 24-Hour Intraocular Pressure (IOP) Profile: Month 12
Description: Response: Yes = had an IOP 24-hour profile; No = did not have an IOP 24-hour profile.
Time Frame: Month 12
Population: PP; N = number of participants with analyzable data at observation.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 436
Participants
  Yes | 60
  No | 376

3. Primary Outcome: Number of Participants With a 24-Hour Intraocular Pressure (IOP) Profile: Month 24
Description: Response: Yes = had an IOP 24-hour profile; No = did not have an IOP 24-hour profile.
Time Frame: Month 24
Population: PP; N = number of participants with analyzable data at observation.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 423
Participants
  Yes | 56
  No | 367

4. Primary Outcome: Number of Participants Per Visit With Intraocular Pressure (IOP) 24-Hour Pressure Peaks: Month 12
Description: Response: Yes = had IOP 24-hour pressure peak; No = did not have IOP 24-hour pressure peak.
Time Frame: Month 12
Population: PP; N = number of participants with analyzable data at observation. The total number of participants by visit with an IOP peak response of 'Yes' differs from those with numerical values of IOP peaks since 1 of the 2 fields was populated for certain participants.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 120
Participants
  Yes | 6
  No | 114

5. Primary Outcome: Number of Participants Per Visit With Intraocular Pressure (IOP) 24-Hour Pressure Peaks: Month 24
Description: Response: Yes = had IOP 24-hour pressure peak; No = did not have IOP 24-hour pressure peak.
Time Frame: Month 24
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 107
Participants
  Yes | 6
  No | 101

6. Primary Outcome: Percentage of Participants Who Achieved Intraocular Pressure (IOP) Target at Last Visit
Description: Percentage of participants who achieved their IOP target set at baseline. Response: Yes = achieved IOP target at last vist; No = did not achieve IOP target at last visit.
Time Frame: Month 24, (or last visit)
Population: PP; n = number of subjects in the Per Protocol Analysis Set with a non-missing response at Last Visit. Last visit = last post-baseline visit at which participant provides a value of IOP.
Measure: Number; unit: Percentage of Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Percentage of Participants
  Yes (n = 264) | 56.3
  No (n = 62) | 13.2

7. Primary Outcome: Change From Baseline by Visit in Optic Disc Excavation: Horizontal Cup to Disc Ratio
Description: Mean horizontal cup to disc (cup/disc or C/D) ratio measured by slit lamp examination to assess progression of glaucoma; calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc). Valid range: 0.1-1.0. Only data for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: PP; N = number of participants with horizontal cup to disc ratio data at baseline and at least 1 post-baseline visit; change analyzed for participants with a non-missing response at baseline and observation. Last Visit: change in participants with a non-missing response at both baseline and at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Xalatan®
Number analyzed (Participants) | 394
Ratio
  Month 6 | -0.00 (0.07)
  Month 12 | 0.00 (0.10)
  Month 18 | 0.01 (0.11)
  Month 24 | 0.01 (0.11)
  Last Visit | 0.00 (0.12)

8. Primary Outcome: Change From Baseline by Visit in Optic Disc Excavation: Vertical Cup to Disc Ratio
Description: Mean vertical cup to disc (cup/disc or C/D) ratio measured by slit lamp examination to assess progression of glaucoma; calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc). Valid range: 0.1-1.0; a high cup/disc ratio may imply glaucoma. Only data for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: PP. N = number of participants with vertical cup to disc ratio at baseline and at least 1 post-baseline visit; change analyzed for participants with a non-missing response at baseline and observation. Last Visit: change in vertical cup to disc ratio in participants with a non-missing response at both baseline and at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Xalatan®
Number analyzed (Participants) | 374
Ratio
  Month 6 | 0.01 (0.08)
  Month 12 | 0.01 (0.10)
  Month 18 | 0.00 (0.11)
  Month 24 | 0.01 (0.11)
  Last Visit | 0.00 (0.12)

9. Primary Outcome: Number of Participants With Optic Disc Hemorrhage by Visit: Month 6
Description: Presence of optic disc hemorrhages assessed by slip lamp examination. Only data for eye were treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Month 6
Population: PP; N = number of participants who indicated whether or not they had an optic disc hemorrhage at the given visit.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 368
Participants | 7

10. Primary Outcome: Number of Participants With Optic Disc Hemorrhage by Visit: Month 12
Description: as for outcome 9
Time Frame: Month 12
Population: PP; N = number of participants who indicated whether or not they had an optic disc hemorrhage at the given visit.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 364
Participants | 6

11. Primary Outcome: Number of Participants With Optic Disc Hemorrhage by Visit: Month 18
Description: as for outcome 9
Time Frame: Month 18
Population: PP; N = number of participants who indicated whether or not they had an optic disc hemorrhage at the given visit.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 373
Participants | 9

12. Primary Outcome: Number of Participants With Optic Disc Hemorrhage by Visit: Month 24
Description: as for outcome 9
Time Frame: Month 24
Population: PP; N = number of participants who indicated whether or not they had an optic disc hemorrhage at the given visit.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 366
Participants | 5

13. Primary Outcome: Change From Baseline in Heidelberg Retina Tomograph (HRT) Parameters: Rim Area
Description: Rim area (millimeter [mm]2) right and left eye assessed by HRT imaging. Valid range: 0.500 to 1.900 mm2. Only the rim area for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: PP; n = number of participants with a non-missing response at both visits (baseline and observation). Last Visit = last post-baseline visit at which participant provides a value for rim area.
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
mm2
  Month 6 (n = 47) | -0.01 (0.11)
  Month 12 (n = 65) | -0.01 (0.15)
  Month 18 (n = 63) | -0.02 (0.17)
  Month 24 (n = 70) | -0.03 (0.16)
  Last Visit (n = 111) | -0.02 (0.16)

14. Primary Outcome: Change From Baseline in Heidelberg Retina Tomograph (HRT) Parameters: Rim Volume
Description: Rim volume (mm3) right and left eye assessed by HRT imaging. Valid range: 0.080 to 0.700 mm3. Only the rim volume for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: PP; n = number of participants with a non-missing response at both visits (baseline and observation). Last Visit = last post-baseline visit at which participant provides a value for rim volume.
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
mm3
  Month 6 (n = 46) | 0.01 (0.06)
  Month 12 (n = 65) | 0.00 (0.06)
  Month 18 (n = 62) | 0.01 (0.11)
  Month 24 (n = 70) | -0.00 (0.05)
  Last Visit (n = 112) | 0.00 (0.08)

15. Primary Outcome: Change From Baseline in Heidelberg Retina Tomograph Parameters: Cup Shape Measure
Description: Cup shape measure right and left eye assessed by HRT imaging . Valid range: -0.400 to -0.010. Only the cup shape measure for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: PP; n = number of participants with a non-missing response at both visits (baseline and observation). Last Visit = last post-baseline visit at which participant provides a value for cup shape measure.
Measure: Mean (Standard Deviation); unit: Cup shape measure
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Cup shape measure
  Month 6 (n = 47) | -0.00 (0.02)
  Month 12 (n = 69) | -0.00 (0.04)
  Month 18 (n = 65) | -0.00 (0.05)
  Month 24 (n = 71) | -0.01 (0.04)
  Last Visit (n = 113) | -0.00 (0.05)

16. Primary Outcome: Change From Baseline in Heidelberg Retina Tomograph (HRT) Parameters: Mean RNFL Thickness
Description: Mean retinal nerve fiber layer (RNFL) thickness in millimeters (mm) right and left eye assessed by HRT imaging. Valid range: 0.100 to 0.400 mm. Only the RNFL for the eye treated with Xalatan® was used; if both eyes were treated, the value of the right eye was analyzed.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24, Last Visit
Population: PP; n = number of participants with a non-missing response at both visits (baseline and observation). Last Visit = last post-baseline visit at which participant provides a value for RNFL thickness.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
mm
  Month 6 (n = 47) | -0.00 (0.03)
  Month 12 (n = 67) | -0.01 (0.04)
  Month 18 (n = 63) | -0.00 (0.05)
  Month 24 (n = 69) | 0.00 (0.04)
  Last Visit (n = 110) | 0.00 (0.05)

17. Primary Outcome: Number of Participants With Change From Baseline to Month 24 in Aulhorn Stages
Description: Values of change in Aulhorn Stage measured by Humphrey Visual Field Analyzer. Aulhorn stages: no scotoma, Stage I (relative scotomas only), Stage II (absolute scotomas without connection to blind spot), Stage III (absolute scotomas with connection to blind spot), Stage IV (absolute scotomas more than 1 quadrant affected), and Stage V (temporal residual visual field only). If both eyes were treated with Xalantan® the value of right eye was analyzed; otherwise, only the assessment for the eye treated with study medication was used.
Time Frame: Baseline, Month 24
Population: PP; N = number of participants who provided Aulhorn stage values of 1 to 5 at both baseline and month 24 visits.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 62
Participants
  Change in Aulhorn Stage: -4 | 1
  Change in Aulhorn Stage: -3 | 2
  Change in Aulhorn Stage: -2 | 0
  Change in Aulhorn Stage: -1 | 6
  Change in Aulhorn Stage: 0 | 45
  Change in Aulhorn Stage: +1 | 6
  Change in Aulhorn Stage: +2 | 2
  Change in Aulhorn Stage: +3 | 0
  Change in Aulhorn Stage: +4 | 0

18. Primary Outcome: Number of Participants With Change From Baseline to Month 24 in Visual Field Defect
Description: Change in mean defect right and left eye; valid range: -30 - + 30 decibels (dB). Visual field defect categories: preperimetric glaucoma: ≥ -2 dB; mild damage: < -2 dB and ≥ -3.3 dB; moderate damage: < -3.3 dB and ≥ -4.6 dB; and severe damage: < -4.6 dB. If both eyes were treated with Xalatan® , the value for the right eye was used; otherwise, only the mean defect value for the eye treated with study medication was used.
Time Frame: Baseline, Month 24
Population: PP; N = number of participants who provided a Mean Defect value at both Baseline and Month 24 visits.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 138
Participants
  Change in mean defect: < 0dB | 60
  Change in mean defect: 0 to < 0.5dB | 31
  Change in mean defect: ≥ 0.5dB to < 1.5dB | 17
  Change in mean defect: ≥ 1.5dB to < 2.5dB | 12
  Change in mean defect: ≥ 2.5dB to < 3.5dB | 6
  Change in mean defect: ≥ 3.5dB to < 4.5dB | 5
  Change in mean defect: ≥ 4.5dB | 7

19. Primary Outcome: Number of Participants With Investigator Assessments of Efficacy at Month 24
Description: Number of participants with Investigator assessments of the efficacy of Xalatan® treatment rated as: 1=very good, 2=good, 3=moderate, 4=insufficient. If study medication was stopped before 24 months, assessment was performed at the time of early termination.
Time Frame: Month 24
Population: PP; N = number of participants with a non-missing response at Month 24 visit.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 442
Participants
  Very Good | 269
  Good | 147
  Moderate | 24
  Insufficient | 2

20. Primary Outcome: Number of Participants With Individual Progression of Glaucoma Damage: Horizontal Cup to Disc Ratio and/or Vertical Cup to Disc Ratio
Description: Increase in Horizontal Cup to Disc Ratio and/or Vertical Cup to Disc Ratio by at least 0.2 (Last Visit minus Baseline).
Time Frame: Month 24 (or last visit)
Population: PP; results based on participants with both a Baseline and at least one post-baseline visit. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Participants | 34

21. Primary Outcome: Number of Participants With Individual Progression of Glaucoma Damage: Optic Disc Hemorrhage
Description: Participants with at least one post-baseline optic disc hemorrhage.
Time Frame: Month 24 (or last visit)
Population: PP; results based on participants with at least one post-baseline assessment of optic disc hemorrhage. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Particpants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Particpants | 16

22. Primary Outcome: Number of Participants With Individual Progression of Glaucoma Damage: Rim Area, Rim Volume, or Mean Retinal Nerve Fiber Layer (RNFL) Thickness
Description: Decrease in at least one Heidelberg Retina Tomograph (HRT) parameter by: Rim Area 0.2 millimeter (mm)2, Rim Volume 0.1 mm3, or mean retinal nerve fiber layer (RNFL) Thickness 0.1 mm, (Last Visit minus Baseline).
Time Frame: Month 24 (or last visit)
Population: PP; results based on participants with a value of the variable in question at both Baseline and at least one post-baseline visit. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Participants | 12

23. Primary Outcome: Number of Participants With Individual Progression of Glaucoma Damage: Visual Field Defect-Deterioration
Description: Visual Field Deterioration rated as progressive by physician on at least one post-baseline visit; range: 1= improved 2= stable 3= progressive. If both eyes were treated with Xalatan® the value for the right eye was used; otherwise, only the assessment for the eye treated with study medication was used.
Time Frame: Month 24 (or last visit)
Population: PP; results based on participants with at least one post-baseline assessment of change in visual field defect. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Participants | 51

24. Primary Outcome: Number of Participants With Individual Progression of Glaucoma Damage: Aulhorn Stage
Description: Increase in Aulhorn Stage by at least one stage (last visit minus baseline). Three different visual field defect categories defined using Aulhorn stage values 1-5: Aulhorn stage 1 = mild damage, Aulhorn stages 2, 3 = moderate damage, Aulhorn stages 4, 5 =severe damage.
Time Frame: Month 24 (or last visit)
Population: PP; results based on participants with a value for Aulhorn Stage at both Baseline and at least one post-baseline visit. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Participants | 20

25. Primary Outcome: Number of Participants With Individual Progression of Glaucoma Damage: Mean Defect
Description: Decrease in mean defect by at least 2.5 decibels (dB) (Last Visit minus Baseline).
Time Frame: Month 24 (or last visit)
Population: PP; results based on participants with a value for mean defect at both Baseline and at least one post-baseline visit. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Participants | 28

26. Primary Outcome: Percentage of Participants With Overall Progression of Glaucoma Damage
Description: Overall progression defined as at least 1 of the 6 individual progression of glaucoma damage measures met: increase in horizontal cup to disc ratio and/or vertical cup to disc ratio by at least 0.2; at least 1 post Baseline (BL) optic-disc hemorrhage; decreased rim area (0.2 mm2), rim volume (0.1 mm3), mean retinal nerve fiber layer (RNFL)(0.1 mm), progressive visual field deterioration, increase in Aulhorn stage (by at least 1 stage), and/or decrease in mean defect by at least 2.5 decibels [dB])
Time Frame: Month 24 (or last visit)
Population: PP; to be included in the percentage, participants must have provided a response for at least one of the six individual progression of glaucoma damage measures. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Percentage of Participants | 25.8

27. Primary Outcome: Percentage of Participants With Progression of Optic Disc Excavation
Description: Progression (Last Visit minus Baseline) defined as increase in horizontal cup to disc ratio and/or vertical cup to disc ratio by at least 0.2, and/or decrease in at least 1 of Heidelberg Retina Tomograph (HRT) parameters (deterioration of rim area 0.2 mm2; deterioration of rim volume 0.1 mm3 deterioration or mean retinal nerve fiber layer (RNFL) thickness 0.1 mm).
Time Frame: Month 24 (or last visit)
Population: PP; to be included in the percentage, participants must have provided a response for at least one of following events: increase in horizontal or vertical cup to disc ratio, or decrease in rim area, rim volume, or mean RNFL thickness. Last Visit = last post-baseline visit at which participant provides a value for the relevant outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Percentage of Participants | 11.3

28. Primary Outcome: Percentage of Participants With Progression of Visual Field
Description: Progression defined as visual field deterioration rated progressive by physician on at least 1 post-baseline visit, and increase in Aulhorn stage (by at least 1 stage) and/or decrease in mean defect by at least 2.5 dB (Last Visit minus Baseline).
Time Frame: Month 24 (or last visit)
Population: PP; to be included in the percentage, participants must have had Visual Field Deterioration rated as progressive by the physician on at least 1 post-baseline visit, and at least one measure of increase in Aulhorn Stage by at least 1 stage, and decrease in Mean Defect by at least 2 dB (last visit minus baseline).
Measure: Number; unit: Percentage of Participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 469
Percentage of Participants | 3.1

ADVERSE EVENTS:
Description: Safety population: all subjects who received at least 1 dose of study medication. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Xalatan®
Serious Adverse Events (participants affected / at risk) | 6/902
Other Adverse Events (participants affected / at risk) | 24/902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xalatan® (N=902)
Myocardial infarction (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Herpes zoster (Infections and infestations) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xalatan® (N=902)
Angina pectoris (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctival irritation (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 3
Conjunctivitis allergic (Eye disorders) | 4
Diplopia (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Ill-defined disorder (General disorders) | 2
Drug hypersensitivity (Immune system disorders) | 2
Hypersensitivity (Immune system disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Dizziness (Nervous system disorders) | 1
Trigeminal nerve paresis (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Cataract operation (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
Outcome measures for this observational non-interventional study were not designated as primary or secondary measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.